CLINICAL TRIAL: NCT01816217
Title: Comparison of Difficult Intubation Rates Using McGrath Mac Video Laryngoscope vs Standard Macintosh Laryngoscope in Critically Ill Patients - a Prospective Interventional Study
Brief Title: Difficult Intubation in Intensive Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The interim analysis has shown a significative difference between the two groups of patients.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UF 8977
Record Dates: First submitted 2013-03-13; First posted 2013-03-22 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Difficult Intubation in ICU; Strictly More Than Two Laryngoscopies; Cormack Grade Three/Four
Keywords: Difficult intubation; Complications; Intensive care units; Videolaryngoscope; Laryngoscopy
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intubated patient (Experimental): Adult intubated in Intensive Care Unit (ICU) with The McGrath Mac videolaryngoscope (intervention described)
  Interventions: Device: Intubation with The McGrath Mac videolaryngoscope

INTERVENTIONS:
Device: Intubation with The McGrath Mac videolaryngoscope

SUMMARY:
Difficult intubation is associated with a worse outcome in intensive care unit (ICU). New videolaryngoscope devices are proposed to improve airway management in ICU patients. We aimed to compare a new videolaryngoscope called " McGrath Mac Video Laryngoscope" vs standard Macintosh Laryngoscope in critically ill patients on difficult intubation and/or Cormack 3-4 rates in a prospective interventional study.The present study was conducted to test the hypothesis that the implementation of a quality-improvement process for airway management using a new videolaryngoscope would be associated with a decreased incidence of difficult intubation and/or Cormack 3-4.

DETAILED DESCRIPTION:
We planned to evaluate in a prospective before-after study performed in a single 16-beds medical-surgical ICU in a teaching hospital that an implementation of a quality-improvement process for airway management using a new videolaryngoscope would be associated with a decreased incidence of difficult intubation and/or Cormack 3-4.During the two periods of the study (non-interventional vs interventional), we planned to evaluate 280 intubations. In the non-interventional phase, all intubations will be performed as the standard of care of the unit using the standard Macintosh laryngoscope for intubation procedure. For this period, 140 intubations will be evaluated and will be considered as a "control" group. After an inter-phase of training on manikin of 6 weeks with the new McGrath mac videolaryngoscope, the "interventional phase will started in aim to include 140 intubations with the McGrath Mac videolaryngoscope.

An intermediate analysis was planned after 70 intubations with McGrath mac videolaryngoscope to assess safety (severe life-threatening complications) and difficult intubation rate and/or Cormack 3-4.Taking into account this intermediate analysis, the number of subjects needed was of 280.

An intubation will be defined as difficult in case of more than two laryngoscopies.

The MACOCHA score and the usual risks factors associated with difficult intubation in operative rooms will be assessed: past difficult intubation, Mallampati score, thyromental distance, mouth opening, neck circumference, upper lip bite test, neck extension, sleep apnea, facial disease.

The following parameters will be recorded: admission diagnosis, age, sex, body mass index, indication for intubation, comorbidities, hour of intubation, SAPS (Simplified Acute Physiologic Score) II score, SOFA (Sequential Organ Failure Assessment) score, skill level of operator,, number of operators, medications used and corresponding doses, equipment used, number of attempts and airway management techniques, head and body position, use of a cricoid pressure.

The complications during intubation will be evaluated:

* respiratory (aspiration, esophageal intubation, saturation less than 80%),
* hemodynamic (systolic arterial pressure less than 65mmHg, high cardiac frequency (more than 150 beats/min) or low cardiac frequency (less than 50 beats/min), arythmias, cardiac arrest),
* neurologic (agitation),
* local (dental injury, airway trauma),
* death.

The complication in the hour following the intubation will be also assessed:

* respiratory: major desaturation (saturation less than 80%, pneumothorax, persistant hypoxia with a saturation less than 80%,
* hemodynamic (persistent hypotension: systolic arterial pressure less than 90mmHg in spite of vascular loading of 500mL of cristalloid solution or 250ml of colloid solution, rythm trouble, cardiac arrest, introduction or increase of vasopressors),
* neurologic (agitation),
* death. Finally, a follow up of 28 days will be done (patient alive at 28 days, or date of death).

ELIGIBILITY:
Inclusion Criteria:

* Patient informed,
* Affiliated or benefit from a disease insurance regimen
* Available for a 28 days follow-up
* Men and women aged aged from at least 18 years
* Indication of intubation in ICU

Exclusion Criteria:

* Protected patient
* Opposition for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The incidence of difficult intubation or/and Cormack 3-4 | during the intubation

SECONDARY OUTCOMES:
The severe life-threatening complications related to intubation in ICU | until 28 days after intubation
  Severe life-threatening complications are defined as death, cardiac arrest, severe cardiovascular collapse, defined as systolic blood pressure<65 mm Hg recorded at least one time and/or <90 mm Hg that lasted 30min despite 500-1,000 ml of fluid loading (crystalloids/or colloids solutions) and/or requiring introduction of vasoactive support, or severe hypoxemia (decrease in SpO2 below 80% during attempts).
The moderate complications related to intubation in ICU | until 28 days after intubation
  Mild to moderate complications are defined as esophageal intubation, aspiration of gastric contents (migration of stomach contents into the lung, supraventricular and/or ventricular arrhythmia (without pulseless rhythm) that require therapy, dangerous agitation (Richmond Agitation-Sedation Scale (RASS) score above 3) or dental injury.
The success rate of intubation on the first attempt | during the intubation
  An intubation attempt is defined as the introduction of the endotracheal tube past the patient's teeth or as a laryngoscopic failure without the introduction of the endotracheal tube. A laryngoscopic blade readjustment counts as a single attempt.
The number of intubation attempts | during the intubation
The glottic view | during the intubation
The success rate | during the intubation

CONTACTS AND LOCATIONS:
Overall Officials: Samir SJ JABER, MD, PhD, Principal Investigator — Anesthesiology and Critical Care Medicine of CHU of Montpellier
Locations (1):
- Centre Hospitalier Universitaire Montpellier, Saint Eloi, Montpellier, Languedoc-Roussillon, France